CLINICAL TRIAL: NCT05472233
Title: The Effect of Sutures Removal Protocols on Coronally Advanced Flap for Root Coverage Outcomes: a Retrospective Study
Brief Title: Effect of Suturing Protocols on Coronally Advanced Flap for Root Coverage Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Nicola Alberto Valente, DDS, MS, PhD, Assistant Professor, University of Cagliari
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Perio1
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recession
Keywords: Gingival recession; Sutures; Root coverage; Healing
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Retrospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2weeks (Active Comparator): Suture removal at 2 weeks post intervention
  Interventions: Procedure: Suture removal after Coronally Positioned Flap
- 3+weeks (Experimental): Suture removal at 3 weeks minimum post intervention
  Interventions: Procedure: Suture removal after Coronally Positioned Flap

INTERVENTIONS:
Procedure: Suture removal after Coronally Positioned Flap — Sutures are removed after different healing period post coronally positioned flap surgery, this latter is a procedure that aims at surgically advancing the gingiva in order to cover dehiscences of the soft tissues uncovering dental roots.

SUMMARY:
The purpose of this retrospective study is to investigate whether suturing protocols (suture removal timing) influence root coverage outcomes in recession defects treated with a coronally advanced flap (CAF) procedure.

DETAILED DESCRIPTION:
The aim of this study is to assess whether the timing of suture removal may influence the number of sites exhibiting complete coverage (CRC) or the mean root coverage (MRC) obtained in single-tooth recession-type defects treated by coronally advanced flap (CAF).

Records from patients that underwent a coronally advanced flap (CAF) procedure for root coverage will be analyzed. This surgical procedure is aimed at the treatment of root recessions that may arise following periodontal disease or mechanical trauma. The procedure, after obtaining deep local anesthesia, involves a sulcular incision on the buccal side and extending the incision mesially and distally to the base of the adjacent papillae. Two vertical incisions are then made at the corner of the adjacent tooth line and extended into the alveolar mucosa. A mixed thickness flap is then elevated and coronally advanced by releasing incisions through the periosteum to allow for flap placement to cover the recession without tension. The papillae are de-epithelized to provide the bed of connective tissue for the adaptation of the flap which is then sutured with single stitches.

The records, complete with photographic documentation, of all patients who have undergone this procedure will be identified and will be divided into two groups: those in which the sutures were removed at 2 weeks and those in which the sutures were removed at 3 or more weeks.

CRC as present or absent (yes/no) and MRC (percentage of roof surface that has been successfully covered) six months after surgery will be assessed in these patients.

The presence of patient discomfort on the day of suture removal will be recorded as present / absent to assess whether the permanence of the sutures for longer or shorter influences the patient's perception of the surgery.

The results will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients not affected by active periodontitis
* Single recessions on non-restored non-molar teeth
* CAF protocols using vertical releasing incisions
* records of patients clearly reporting timing of suture removals and root coverage outcomes at 6 months

Exclusion Criteria:

* Adjacent recessions
* Recessions on molar teeth
* Coronally advanced flaps without releasing incisions
* Patients with active periodontitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Complete Root Coverage | 6 months
  Achievement of 100% root coverage, measured as yes / no
Mean Root Coverage | 6 months
  Percentage of the root recession that has been successfully covered after the surgical procedure

SECONDARY OUTCOMES:
Patient discomfort | at suture removal
  Discomfort reported by the patient (present/absent)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Duilio Casula, AOU Cagliari, Monserrato, CA, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared in a publication after the end of the study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be submitted for publication right after the analysis of the outcomes

REFERENCES:
- [Background] Tatakis DN, Chambrone L. The Effect of Suturing Protocols on Coronally Advanced Flap Root-Coverage Outcomes: A Meta-Analysis. J Periodontol. 2016 Feb;87(2):148-55. doi: 10.1902/jop.2015.150394. Epub 2015 Oct 8. PMID 26447751
- [Background] Tavelli L, Barootchi S, Ravida A, Suarez-Lopez Del Amo F, Rasperini G, Wang HL. Influence of suturing technique on marginal flap stability following coronally advanced flap: a cadaver study. Clin Oral Investig. 2019 Apr;23(4):1641-1651. doi: 10.1007/s00784-018-2597-5. Epub 2018 Aug 27. PMID 30151706
- [Background] Huang LH, Wang HL. Sling and tag suturing technique for coronally advanced flap. Int J Periodontics Restorative Dent. 2007 Aug;27(4):379-85. PMID 17726994
- [Background] Huang LH, Neiva RE, Wang HL. Factors affecting the outcomes of coronally advanced flap root coverage procedure. J Periodontol. 2005 Oct;76(10):1729-34. doi: 10.1902/jop.2005.76.10.1729. PMID 16253095
- [Background] Tatakis DN, Chambrone L, Allen EP, Langer B, McGuire MK, Richardson CR, Zabalegui I, Zadeh HH. Periodontal soft tissue root coverage procedures: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S52-5. doi: 10.1902/jop.2015.140376. Epub 2014 Oct 15. PMID 25315018
- [Background] Chambrone L, Pannuti CM, Tu YK, Chambrone LA. Evidence-based periodontal plastic surgery. II. An individual data meta-analysis for evaluating factors in achieving complete root coverage. J Periodontol. 2012 Apr;83(4):477-90. doi: 10.1902/jop.2011.110382. Epub 2011 Aug 22. PMID 21859324